CLINICAL TRIAL: NCT01944215
Title: Evaluation of the Effect of Fasting and Exercise on Uptake of Tc-99m Sestamibi in Breast Tissue
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael O'Connor, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-004749; R44CA143716 (NIH)
Record Dates: First submitted 2013-09-04; First posted 2013-09-17 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2015-12

CONDITIONS: Molecular Imaging
Keywords: Normal subjects; Female; Molecular Breast Imaging; Fasting; Exercise; Tracer Uptake; Tc-99m Sestamibi; Prandial status; metabolic status; negative mammogram; Caffeine; External Warming
MeSH Terms: conditions — Fasting; Motor Activity | interventions — Meals; Exercise; Technetium Tc 99m Sestamibi; Technetium; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 4 - Fast vs Fast + External Heating (Active Comparator): MBI will be performed in 52 subjects after an overnight fast with 4-6 mCi Tc-99m sestamibi. The subject will receive the usual Mayo gown for breast imaging. A skin temperature sensor will be taped to the anterior of one breast and skin temperature will be recorded. The subject will be asked to sit for 15 minutes in the waiting room prior to injection of the Tc-99m sestamibi. Just prior to injection, skin temperature will be recorded again. After completion of the first study the subject will then be given a warm towel robe and a small heating pad to be placed over the chest area. After 30 minutes, skin temperature will be recorded again immediately prior to injection of the second dose of Tc-99m sestamibi. The second MBI study will then be performed.
  Interventions: Radiation: Sestamibi; Other: External Heating
- Arm 3 - Fasting vs. Fasting + Caffeine (Active Comparator): MBI will be performed in 52 subjects after an overnight fast with 4-6 mCi Tc-99m sestamibi. The subject will then be instructed to consume 200 mg caffeine in tablet form. This is equivalent to the caffeine content of an 8 oz brewed coffee from Starbucks. After 45 minutes after consumption of the caffeine tablet, patients will receive a second injection of 4-6 mCi Tc-99m sestamibi and a repeat MBI study will be performed.
  Interventions: Radiation: Sestamibi; Drug: Caffeine Tablet
- Arm 2-Resting vs. Exercising (Active Comparator): MBI will be performed in 25 subjects after an overnight fast with 4-6 mCi Tc-99m sestamibi. Patients will then be asked to perform moderate exercise on a treadmill for 6-10 minutes at a level of 70%-80% of maximum predicted heart rate. At ~10 minutes, patients will receive a second injection of 4-6 mCi Tc-99m sestamibi and a repeat MBI study will be performed.
  Interventions: Other: Exercise; Radiation: Sestamibi
- Arm 1-Fasting vs. Fed (Active Comparator): MBI will be performed in 25 subjects after an overnight fast with 4-6 mCi Tc-99m sestamibi. Patients will then be instructed to consume 8-16 fluid oz of Ensure (350-700 calories). At 30 minutes after consumption of the meal, patients will receive a second injection of 4-6 mCi Tc-99m sestamibi and a repeat MBI study will be performed.
  Interventions: Dietary Supplement: Meal; Radiation: Sestamibi

INTERVENTIONS:
Dietary Supplement: Meal — effect of meal
  Other Names: Ensure
  Arms: Arm 1-Fasting vs. Fed
Other: Exercise — effect of exercise
  Arms: Arm 2-Resting vs. Exercising
Radiation: Sestamibi — reduce radiation dose
  Other Names: Tc-99m
Drug: Caffeine Tablet — effect of caffeine
  Other Names: 200 mg Vivarin Tablet
  Arms: Arm 3 - Fasting vs. Fasting + Caffeine
Other: External Heating — Heating Pad and warm blanket robe
  Arms: Arm 4 - Fast vs Fast + External Heating

SUMMARY:
The primary objective of this study is to determine if exercise, fasting, or eating prior to the molecular breast imaging study will have an effect on the uptake of the tracer in the breast tissue.

DETAILED DESCRIPTION:
The primary objective of this study is to determine if exercise, fasting, or eating prior to a molecular breast imaging study will have an effect on the uptake of the radiotracer Tc-99m sestamibi in the breast tissue.

Tc-99m sestamibi is primarily extracted by the liver. Changes in hepatic blood flow may therefore influence the amount of radiotracer available for uptake in the breast tissue.

ELIGIBILITY:
Inclusion criteria:

Arm 1: 1. Able to fast overnight or for 6 hours 2. Non-diabetic 3. Age > 40 years 4. Negative pregnancy test, postmenopausal, or surgically sterilized 5. Negative mammogram at Mayo Clinic within the last 15 months (defined as screening mammogram or subsequent diagnostic workup with BI-RADS 1 or 2 final assessment) 6.No current breast concerns

Arm 2: 1. Able to fast overnight or for 6 hours 2. Able to perform light to moderate exercise on an exercise bike 3. Non-diabetic and Body Mass Index < 25 4. Age > 40 years and < 70 years 5. Negative pregnancy test, postmenopausal, or surgically sterilized 6. Negative mammogram at Mayo Clinic within the last 15 months (defined as screening mammogram or subsequent diagnostic workup with BI-RADS 1 or 2 final assessment) 7. No current breast concerns 8. No history of coronary artery disease, angina, stroke or peripheral arterial disease.

Arm 3: 1. Able to fast overnight or for 6 hours 2. Willing to consume a dose of caffeine (200 mg), equivalent to that of an 8 oz Starbuck brewed coffee.

3. Non-diabetic 4. Age > 40 years 5. Negative pregnancy test, postmenopausal, or surgically sterilized 6. Negative mammogram at Mayo Clinic within the last 15 months (defined as screening mammogram or subsequent diagnostic workup with BI-RADS 1 or 2 final assessment) 7. No current breast concerns

Arm 4: 1. Able to fast overnight or for 6 hours 2. Non-diabetic 3. Age > 40 years 4. Negative pregnancy test, postmenopausal, or surgically sterilized 5. Negative mammogram at Mayo Clinic within the last 15 months (defined as screening mammogram or subsequent diagnostic workup with BI-RADS 1 or 2 final assessment) 6. No current breast concerns

Exclusion Criteria:

* Pregnancy test (if necessary) is not negative, or the patient is unable to complete the pregnancy test
* Physically unable to sit upright and still remain still during two consecutive MBI studies over the course of a 2 hour period.
* Have undergone unilateral or bilateral mastectomy
* Breast implants or silicone injections
* Are unable to understand and sign the consent form
* Arm 2-also includes: Unable to perform light to moderate exercise for 12 minutes on a treadmill or a stationary bicycle
* Arm 3: Unwilling to consume a 200 mg dose of caffeine

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Uptake of this radiopharmaceutical in breast tissue | 2 Days
  Quantitative measurements of Tc-99m sestamibi uptake will be performed to measure the relative change in uptake between the two MBI scans.

CONTACTS AND LOCATIONS:
Overall Officials: Michael K O'Connor, PhD, R-D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Rhodes DJ, Hruska CB, Phillips SW, Whaley DH, O'Connor MK. Dedicated dual-head gamma imaging for breast cancer screening in women with mammographically dense breasts. Radiology. 2011 Jan;258(1):106-18. doi: 10.1148/radiol.10100625. Epub 2010 Nov 2. PMID 21045179
- [Derived] Swanson TN, Tran TD, Hruska CB, Solberg CM, Rhodes DJ, Hunt KN, Conners AL, O'Connor MK. Patient Acceptance of Half-dose Vs. Half-time Molecular Breast Imaging. J Med Imaging Radiat Sci. 2018 Mar;49(1):39-43. doi: 10.1016/j.jmir.2017.08.003. Epub 2017 Sep 13. PMID 30479286
- [Derived] O'Connor MK, Hruska CB, Tran TD, Swanson T, Conners AL, Jones K, Rhodes DJ. Factors influencing the uptake of 99mTc-sestamibi in breast tissue on molecular breast imaging. J Nucl Med Technol. 2015 Mar;43(1):13-20. doi: 10.2967/jnmt.114.150128. Epub 2015 Jan 22. PMID 25613340
- See also: Molecular Breast Imaging-Mayo Clinic — http://www.youtube.com/watch?v=DOQBLe8MdH0